CLINICAL TRIAL: NCT02039492
Title: Sympathetic Renal Denervation Versus Increment of Pharmacological Treatment in Resistant Arterial Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Anna Oliveras, PhD, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DENERVHTA
Record Dates: First submitted 2014-01-16; First posted 2014-01-17 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Resistant Arterial Hypertension
MeSH Terms: interventions — Therapeutics; Spironolactone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Denervation
  Interventions: Procedure: Sympathetic Renal Denervation
- B (Active Comparator): Treatment with aldactone
  Interventions: Drug: Treatment with aldactone

INTERVENTIONS:
Procedure: Sympathetic Renal Denervation
  Arms: A
Drug: Treatment with aldactone
  Arms: B

SUMMARY:
Background: In hypertension, a highly prevalent disease, up to 10-15% of hypertensive patients have uncontrolled blood pressure despite a regimen of ≥ 3 drugs, which is known as resistant hypertension (RH). Cardiovascular prognosis in patients with RH is worse than in controlled hypertensives. Efferent renal sympathetic nerves play an important role in volume homeostasis and blood pressure. A novel minimally invasive technique based on the use of selective radiofrequency renal sympathetic denervation has shown promising preliminary results for the treatment of these patients. On the other hand, some patients with RH could improve their blood pressure control by adding spironolactone, an antagonist of aldosterone receptors.

Objective: To evaluate the efficacy of radiofrequency renal sympathetic denervation in patients with RH, as compared with the addition of spironolactone to the therapeutic regimen at baseline.

Method: interventional, prospective, randomized, open study, of a cohort of 50 patients with RH, with office systolic blood pressure ≥ 150 mmHg and also with 24h systolic blood pressure ≥ 140 mmHg, despite treatment with ≥ 3 drugs in adequate doses, one of them a diuretic, and whitout treatment with either spironolactone or eplerenone. Patients will be randomized (1:1) to renal sympathetic denervation treatment or spironolactone (50mg), performing determination of office blood pressure and 24h-ABPM at pre-randomization, 1, 3 and 6 months, as well as laboratory tests, echocardiography, measurement of carotid intima-media thickness and central blood pressure measurement at pre-randomization and after 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged ≥ 18 years and ≤ 80 years.
2. Subjects with diagnosed resistant arterial hypertension (office blood pressure ≥ 140 and/or 90 mm Hg despite treatment with at least 3 antihypertensive drugs given at the maximum tolerated therapeutic dosage, being one of them a diuretic), with this therapeutic regimen maintained for at least the last 3 months.
3. Office systolic blood pressure ≥150 mm Hg, with confirmation of resistance to treatment by 24h ambulatory blood pressure monitoring, with 24h-systolic blood pressure ≥140 mmHg being required to be included.
4. Patients who have freely given informed consent in writing, after the nature of the study and the disclosure of their data have been explained to them.

Exclusion Criteria:

* 1. Secondary hypertension, renovascular disease included with appropriate tests according to investigator criteria (with the exceptions of chronic renal disease and obstructive sleep-apnea syndrome). 2. Inability to perform magnetic resonance angiography or renal CT angiography (contrast allergy). 3. Patients unlikely compliant with treatment (assessed according to Haynes-Sackett test). 4. Patients currently on treatment with an aldosterone receptor blocker (spironolactone, eplerenone) or who had previously received one of such class of drugs and had been withdrawn due to lack of efficacy and/or adverse effects. 5. Stage 3B, 4 or 5 of chronic renal disease (estimated glomerular filtration rate by MDRD equation < 45 mL/min/1.73m2). 6. Pre-randomization serum potassium (K+) level ≥ 5.5 mmol/L. 7. Significant renal vascular anomalies. 8. Pregnant women. 9. Significant valvular heart disease. 10. Major vascular event (myocardial infarction, unstable angina or cerebrovascular disease) < 6 months prior to study enrolment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Changes in ambulatory 24h-systolic blood pressure (SBP). | From baseline (Visit 0) to Final Examination (6 months).

SECONDARY OUTCOMES:
Changes in ambulatory 24h-diastolic blood pressure (DBP), pulse pressure (PP) and heart rate (HR) | From baseline (Visit 0) to Final Examination (6 months).

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital General de l'Hospitalet, Hospitalet, Barcelona
  - Hospital Universitari Mútua de Terrassa, Terrassa, Barcelona

REFERENCES:
- [Derived] Oliveras A, Armario P, Sans L, Clara A, Vazquez S, Molina L, Pareja J, de la Sierra A, Pascual J. Organ damage changes in patients with resistant hypertension randomized to renal denervation or spironolactone: The DENERVHTA (Denervacion en Hipertension Arterial) study. J Clin Hypertens (Greenwich). 2018 Jan;20(1):69-75. doi: 10.1111/jch.13156. Epub 2018 Jan 5. PMID 29316186
- [Derived] Oliveras A, Armario P, Clara A, Sans-Atxer L, Vazquez S, Pascual J, De la Sierra A. Spironolactone versus sympathetic renal denervation to treat true resistant hypertension: results from the DENERVHTA study - a randomized controlled trial. J Hypertens. 2016 Sep;34(9):1863-71. doi: 10.1097/HJH.0000000000001025. PMID 27327441